CLINICAL TRIAL: NCT06963320
Title: A Multicenter, Randomized, Open-label, Positive-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of H001 Capsules in the Prevention of Venous Thromboembolism (VTE) in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Phase II Clinical Study of H001 Capsule in the Prevention of Venous Thromboembolism After Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LZ-033-II
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Circulatory Disease
MeSH Terms: interventions — enoxaparin sodium; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- H001 Capsule 200mg-qd (Experimental)
  Interventions: Drug: H001 Capsule 200mg-qd
- H001 Capsule 300mg-qd (Experimental)
  Interventions: Drug: H001 Capsule 300mg-qd
- H001 Capsule 200mg-bid (Experimental)
  Interventions: Drug: H001 Capsule 200mg-bid
- Enoxaparin Sodium Injection (Active Comparator)
  Interventions: Drug: Enoxaparin Sodium Injection

INTERVENTIONS:
Drug: H001 Capsule 200mg-qd — H001 Capsule, 50 mg/capsule, 200 mg orally once daily for 10-14 days.
  Arms: H001 Capsule 200mg-qd
Drug: Enoxaparin Sodium Injection — Enoxaparin Sodium Injection,0.4 mL: 4000 AXaIU, 40 mg subcutaneously once daily for 10-14 days
  Arms: Enoxaparin Sodium Injection
Drug: H001 Capsule 300mg-qd — H001 Capsule, 50 mg/capsule, 300 mg orally once daily for 10-14 days.
  Arms: H001 Capsule 300mg-qd
Drug: H001 Capsule 200mg-bid — H001 Capsule, 50 mg/capsule, 200 mg orally twice daily for 10-14 days.
  Arms: H001 Capsule 200mg-bid

SUMMARY:
This study is a multicenter, randomized, open-label, positive-controlled Phase II clinical study to evaluate the efficacy and safety of H001 capsules in the prevention of venous thromboembolism (VTE) in subjects undergoing Total Knee Arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo elective primary unilateral total knee arthroplasty (TKA);
2. Aged 18-74 years (inclusive) on the day of signing the informed consent form, regardless of gender;
3. Willing and able to voluntarily sign the informed consent form and comply with the study protocol;
4. Women of childbearing potential or subjects whose partners are women of childbearing potential must agree to use effective contraception throughout the study period. Acceptable methods include oral, implantable, or injectable hormonal contraceptives; mechanical products (e.g., intrauterine devices, diaphragms, condoms, spermicides); abstinence; or confirmed sterilization (e.g., vasectomy, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Exclusion Criteria:

1. Pregnant or breastfeeding female subjects;
2. Body weight <40 kg at screening;
3. History of allergy to contrast agents or inability to undergo bilateral lower limb venography; history of hypersensitivity to the study drug or drugs of the same class; known allergy to enoxaparin or any component listed in the enoxaparin prescribing information;
4. High bleeding risk or contraindications to enoxaparin (e.g., known or suspected heparin-induced thrombocytopenia, severe hematologic disorders, severe coagulation abnormalities);
5. History of deep vein thrombosis (DVT) or DVT confirmed during screening;
6. Clinically significant medical history, including

   1. Hemorrhagic stroke or intracranial conditions (e.g., hemorrhage, tumor, arteriovenous malformation, or aneurysm);
   2. Recurrent upper gastrointestinal or genital/urinary tract ulcers/bleeding, intraocular bleeding, or clinical bleeding within 6 months prior to screening (as judged by the investigator to increase bleeding risk);
   3. Acute hepatitis within 1 year prior to screening or persistent severe liver disease (e.g., chronic active hepatitis, cirrhosis, or chronic hepatic insufficiency);
   4. Myocardial infarction, acute coronary syndrome, viral myocarditis, pulmonary embolism, or coronary revascularization within 6 months prior to screening; transient ischemic attack or ischemic stroke;
   5. Chronic congestive heart failure with NYHA Class IV cardiac function;
   6. Severe arrhythmias requiring Class Ia or III antiarrhythmic drugs; sinus node dysfunction, Type II Mobitz or third-degree atrioventricular block without pacemaker implantation;
   7. History of QTc interval prolongation or QTc interval ≥480 ms during screening;
7. Poorly controlled hypertension within 3 months prior to screening (defined as failure to achieve target blood pressure despite ≥3 antihypertensive medications) or systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg confirmed during screening;
8. Major surgery or trauma within 3 months prior to screening, particularly involving the brain, spine, or eyes;
9. Use of the following treatments:

   1. Ongoing or recent (within 7 days pre-surgery) anticoagulant therapy (e.g., after mechanical heart valve replacement) or plans to continue such therapy during the study;
   2. Oral antiplatelet therapy (e.g., aspirin >165 mg/day, clopidogrel, ticlopidine, dipyridamole) within 7 days pre-surgery or plans to continue during the study;
   3. Long-acting NSAIDs within 7 days or 5 half-lives (whichever is longer) prior to surgery;
   4. Thrombolytic therapy for ischemic disease within 6 months prior to screening;
10. Planned or ongoing use of epidural analgesia post-surgery; planned or ongoing use of intermittent pneumatic compression devices, electrical/mechanical muscle stimulators post-surgery; intraoperative complications (e.g., hemorrhage or severe trauma) during spinal/epidural anesthesia;
11. Laboratory abnormalities at screening:

    1. Total bilirubin >1.5×ULN, ALT or AST >3×ULN;
    2. Serum creatinine >1.5×ULN; chronic kidney disease with eGFR <30 mL/min/1.73 m²;
    3. Hemoglobin <100 g/L;
    4. Platelet count <100×10⁹/L;
    5. APTT, PT, or INR >ULN with clinical significance (investigator judgment);
12. History of malignancy within 5 years prior to screening (excluding basal cell carcinoma or Stage I squamous cell carcinoma);
13. Positive serum pregnancy test (hCG) during screening;
14. Participation in another drug/device clinical trial within 1 month prior to screening or within 5 half-lives of the investigational drug (whichever is longer);
15. History of drug abuse or psychiatric disorders;
16. Other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of total VTE | Within 14 days post-dose

SECONDARY OUTCOMES:
Major bleeding and clinically relevant non-major bleeding | Within 14 days post-dose
Incidence of total DVT | Within 14 days post-dose
Incidence of Proximal DVT | Within 14 days post-dose
Incidence of Distal DVT | Within 14 days post-dose
Incidence of Total VTE | Within 42 days post-dose
Major bleeding | Within 42 days post-dose
Clinically relevant non-major bleeding | Within 42 days post-dose
Other bleeding events | Within 42 days post-dose
TEAEs, laboratory tests, ECG, vital signs, physical examination, etc. | Within 42 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China